CLINICAL TRIAL: NCT03771768
Title: Active Control,Randomized,Double- Blinded Clinical Trial of BD
Brief Title: Diode Laser Versus Topical Corticosteroids in Management of Oral Ulcers in Behcet's Disease
Acronym: BD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Clair Sobhy Nagieb Botros, Principal invistigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3:5:1
Record Dates: First submitted 2018-12-01; First posted 2018-12-11 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-02

CONDITIONS: Autoimmune; Behcet Syndrome
Keywords: Oral ulcers
MeSH Terms: conditions — Behcet Syndrome; Oral Ulcer | interventions — Low-Level Light Therapy; Triamcinolone Acetonide; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Care Provider, Investigator
Masking Description: Double - blinded trial:
  Outcome assessor (CS) and Statistician. Participants couldn't be blinded because of the difference in the nature of interventions method of application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triamcinolone acetonide (Active Comparator): Triamcinolone acetonide 0.1% 5 gm adhesive paste 4 times / day for 1 month.
  Interventions: Drug: Triamcinolone Acetonide
- Diode laser (Experimental): Diode laser 980 nm & 100mWatt.
  Interventions: Radiation: Diode laser 980nm&100 mWatt

INTERVENTIONS:
Radiation: Diode laser 980nm&100 mWatt — Diode laser 980 nm &100 milli Watt.
  Other Names: Low level laser; Biostimulation; Soft laser
  Arms: Diode laser
Drug: Triamcinolone Acetonide — 0.1 &5gm paste 4 times/day
  Other Names: Topical corticosteroid
  Arms: Triamcinolone acetonide

SUMMARY:
Laser therapy is increasingly showing promising results in dental field including oral ulcers.This trial will assess the usefulness of Diode Laser compared to corticosteroid on oral ulcers of patients diagnosed with Behcet's disease.

DETAILED DESCRIPTION:
The enrolled patients will be divided randomly into two groups.one group will receive Diode Laser (power:100 milli Watt,wavelength:980 mmm, delivery system:biostimulation probe) and other group will receive topical corticosteroids(Kenacort A Orabase: triamcinolone acetonide 0.1% 5 gram adhesive paste - Dermaphor) four times daily.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Behcet's Disease according to International Criteria for BD.
* patients with active oral ulcers.
* patients free from any visible oral lesions other than the oral ulcers of BD.
* patients who agreed to take the supplied interventions.
* patients who will agree to participate in the study.
* patients who will accept to sign the informed consent.

Exclusion Criteria:

* patients not physically able to participate in survey or clinical oral examination.
* patients with organ or life-threatening disease.
* patients with history of a severe or chronic medical condition including tuberculosis, hepatitis and human immunodeficiency virus.
* patients under immunosuppressive drugs.
* patients with organ transplantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-05-25 (Estimated); Primary Completion 2019-05-25 (Estimated); Study Completion 2019-05-25 (Estimated)

PRIMARY OUTCOMES:
Oral ulcer activity index | One month
  Composite index score (0-10)

SECONDARY OUTCOMES:
Oral health - related quality of life | One month
  Oral health impact profile - 14 (OHIP- 14)
Pain associated with oral ulcer | One month
  Visual analogue scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Sherin Ali Hassan, MD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prasad R S, Pai A. Assessment of immediate pain relief with laser treatment in recurrent aphthous stomatitis. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Aug;116(2):189-93. doi: 10.1016/j.oooo.2013.02.011. Epub 2013 Apr 23. PMID 23622766
- [Background] Hatemi G, Merkel PA, Hamuryudan V, Boers M, Direskeneli H, Aydin SZ, Yazici H. Outcome measures used in clinical trials for Behcet syndrome: a systematic review. J Rheumatol. 2014 Mar;41(3):599-612. doi: 10.3899/jrheum.131249. Epub 2014 Feb 1. PMID 24488418
- [Derived] Nagieb CS, Harhash TA, Fayed HL, Ali S. Evaluation of diode laser versus topical corticosteroid in management of Behcet's disease-associated oral ulcers: a randomized clinical trial. Clin Oral Investig. 2022 Jan;26(1):697-704. doi: 10.1007/s00784-021-04047-8. Epub 2021 Jul 2. PMID 34212234